CLINICAL TRIAL: NCT01810276
Title: The Safety and Efficacy of Platelet Transfusion in Patients Receiving Antiplatelet Therapy That Sustain Traumatic Intracranial Hemorrhage
Brief Title: Safety of Platelet Transfusion in Patients on Antiplatelet Therapy With Traumatic Head Injury
Acronym: PUNCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient population not available
Sponsor: Christiana Care Health Services (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 601291; 31115 (Other: Christiana Care Health System)
Record Dates: First submitted 2012-11-07; First posted 2013-03-13 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Traumatic Head Injury; Intracranial Hemmorhage; Anti-platelet Therapy
Keywords: traumatic head injury; intracranial hemorrhage; platelets; anti-platelet therapy; plavix; asprin
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Sodium Chloride; Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): 400 mL of Saline will be given intravenously over 2 hours once.
  Interventions: Other: Saline
- Platelets (Active Comparator): 2 apheresis units of platelets (approximately 200 ml) will be given intravenously over 2 hours.
  Interventions: Other: Platelets

INTERVENTIONS:
Other: Saline — 400 mL of Saline will be given intravenously over 2 hours once
  Arms: Saline
Other: Platelets — 2 apheresis units of platelets (approximately 200 ml) will be given intravenously over 2 hours.
  Arms: Platelets

SUMMARY:
The objective of this study is to determine if the administration of platelets will improve outcome in patients with ICH who are being treated with either aspirin, a thienopyridine (ticlodipine, clopidogrel, prasugrel) or a combination of both. The study has four specific aims:

1. To determine what affect platelet administration will have on bleeding in the brain.
2. To determine what affect platelet administration will have on brain function. Several assessments to test the functioning of the brain will be performed at enrollment and throughout the study. Comparing the results of these assessments between the experimental and control groups should allow us to determine if platelet administration improves outcomes in patients with bleeding in the brain exposed to antiplatelet therapy.
3. An important risk of reversing antiplatelet therapy is exposing the patient to the very complications this therapy was designed to prevent. Therefore, tracking complications will be a very important part of this study. The investigators will compare the rates of death, heart attack, stroke and clots in the veins between groups.
4. Some patients (10-40%) have limited responsiveness to antiplatelet therapy. While platelet responsiveness, as measured by a special platelet blood test, will not affect enrollment, the investigators feel it will be important to measure.

DETAILED DESCRIPTION:
Intracranial hemorrhage (ICH), or bleeding in the brain, is the major cause of death in trauma patients. The initial volume and early growth of the hematoma are critical determinants of mortality and functional outcome. As our population ages, a significant and growing number of patients present with ICH while on antiplatelet therapy. Bleeding is a well known complication of this therapy. It is likely that patients with ICH who are exposed to antiplatelet therapy would have an increased risk of hemorrhage growth and poor outcome compared to patients that are not using antiplatelet therapy. There are no pharmacologic agents that can reverse the antithrombotic effect of aspirin or the thienopyridines. There is a paucity of published data, one small phase one trial and two retrospective studies that address the use of platelets as a means to reverse the effects of antiplatelet therapy in patients suffering ICH. In addition, transfusion of platelets may be associated with transfusion reactions, such as infection and fluid overload. Furthermore, these patients are then exposed to the very thromboembolic complications the antiplatelet therapy was designed to prevent.

Given the lack of data, which is primarily retrospective and likely underpowered, The investigators feel it's important to conduct a trial to more definitively study the efficacy of antiplatelet reversal in patients with life threatening ICH. Furthermore, it would be important to understand that, if there is a benefit to antiplatelet reversal in patients with ICH, that this benefit will outweigh the risks of antiplatelet reversal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Evidence of intracranial hemorrhage (bleeding in the brain) by CT scan related to traumatic injury
* Receiving antiplatelet therapy such as aspirin, thienopyridine (ticlopidine, clopidogrel, or prasugrel)
* Platelet count greater than or equal to 100,000

Exclusion Criteria:

* Glasgow Coma Scale (GCS) less than 6
* Hemorrhage requiring emergent surgery
* Lack of permission from treating physician and/or consultant
* Secondary ICH related to aneurysm or arteriovenous malformation
* Use of oral anticoagulants
* Decreased platelets (thrombocytopenia)
* Patients requiring massive transfusion protocol
* Life expectancy less than 3 months
* Confirmed acute heart attack
* Hepatitis and liver cirrhosis
* Kidney failure
* Participation in another treatment study within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Hemorrhage growth | 24 hours
  Bleeding in the brain will be measured by computerized tomography scan (CT Scan) 24 hours after study treatment is completed.

SECONDARY OUTCOMES:
Neurological Outcome | Assessments to determine brain function or neurological outcome will be performed at enrollment, time of study treatment, 1 and 24 hours post treatment, days 2, 3, and 10 (or time of discharge) and at 90 days post treatment.
  Assessments to determine brain function or neurological outcome will be performed at enrollment, time of study treatment, 1 and 24 hours post treatment, days 2, 3, and 10 (or time of discharge) and at 90 days post treatment.

OTHER OUTCOMES:
Thromboembolic complications | Complications will be monitored enrollment, time of study treatment, 1 and 24 hours post treatment, days 2, 3, and 10 (or time of discharge)and at 90 days post treatment.
  Complications such as heart attack, stroke, venous thromboembolic, and death which can be caused by reversing antiplatelet therapy will be monitored enrollment, time of study treatment, 1 and 24 hours post treatment, days 2, 3, and 10 (or time of discharge)and at 90 days post treatment.
Platelet responsiveness | 1 hour and 24 hours post study treatment
  Platelet responsiveness will be measured by lab test at 1 and 24 hours post study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cipolle, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Christiana Hospital, Newark, Delaware, United States